CLINICAL TRIAL: NCT01804387
Title: Comparison of Telbivudine Plus Adefovir With Lamivudine Plus Adefovir for the Treatment of Lamivudine-resistant Chronic Hepatitis B at 52 Weeks: A Pilot Study
Acronym: TeSLA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea University (Other)
Responsible Party: Principal Investigator, Hyung Joon Yim, Associate professor, Korea University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TeSLA study
Record Dates: First submitted 2011-12-23; First posted 2013-03-05 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic Hepatitis B; Telbivudine; Adefovir; Lamivudine resistance
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Telbivudine; adefovir; adefovir dipivoxil; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telbivudine plus adefovir (Active Comparator): study drugs
  Interventions: Drug: telbivudine plus adefovir
- Lamivudine plus adefovir (Active Comparator): standard drugs
  Interventions: Drug: lamivudine plus adefovir

INTERVENTIONS:
Drug: telbivudine plus adefovir — telbivudine 600 mg qd plus adefovir 10 mg qd
  Other Names: telbivudine (sevibo); adefovir (hepsera)
  Arms: Telbivudine plus adefovir
Drug: lamivudine plus adefovir — lamivudine 100 mg qd plus adefovir 10mg qd
  Other Names: lamivudine (zeffix); adefovir (hepsera)
  Arms: Lamivudine plus adefovir

SUMMARY:
Lamivudine had been widely used for treatment-naïve chronic hepatitis B patients. However, development of antiviral resistance has been known as the major drawback: Incidence of lamivudine resistance was reported to be approximately 70% after 5 years (Lok AS et al, 2003). For the treatment of lamivudine resistance, adefovir has been widely used (Lok AS and McMahon B, 2009). However, switching to adefovir monotherapy was also reported to be at high risk of resistance, 25% at year 2 (Yeon JE et al, 2006). Recently, adding adefovir on lamivudine was shown to be superior to switching to adefovir monotherapy by decreasing the adefovir resistance (Rapti I et al, 2007, Lampertico P et al, 2007). However, combination of adefovir and lamivudine does not increase antiviral activity compared with adefovir monotherapy in patients with lamivudine resistance (Peters MG et al, 2004). As many patients are still viremic with the treatment of lamivudine and adefovir over 1 year, the investigators need more potent combination of the drugs. Telbivudine is a new nucleoside analogue with potent antiviral activity. The previous phase III study has shown the superiority of telbivudine over lamivudine in HBeAg positive and negative subjects (Lai CL et al, 2007). Therefore, telbivudine plus adefovir may be a better treatment option than lamivudine plus adefovir for the lamivudine-resistant chronic hepatitis B patients. No study assessing the efficacy of telbivudine plus adefovir has been conducted for these patients. The aim of this study is to evaluate the safety and efficacy of telbivudine plus adefovir compared with lamivudine plus adefovir in lamivudine resistant chronic hepatitis B patients at the end of 1 year follow-up,

ELIGIBILITY:
Inclusion Criteria:

1. HBeAg positive or negative chronic hepatitis B patients (positive HBsAg more than 6 months)
2. Age ≥ 18 years old, and ≤70 years old
3. Previous treatment with lamivudine more than 6 months
4. Being on lamivudine at the time of screening
5. Confirmed genotypic resistance to lamivudine by RFMP (rtM204V or I)
6. Presence of virologic breakthrough ≥1 log increase of HBV DNA above na dir)
7. HBV DNA ≥ 20,000 IU/mL
8. Patient willing to give an informed consent (If patient is <20 years old, the parent or legal guardian also need to give an informed consent)

Exclusion Criteria:

1. Out of inclusion criteria
2. Presence of adefovir resistance (rtA181T or V, rtN236T) by RFMP assay
3. Laboratory abnormalities as follows at screening: AFP>100 ng/mL, serum phosphorous level<2.4 mg/dL, serum creatinine level> 1.5 mg/dL or creatinine clearance < 50 mL/min
4. Patient with a history of decompensated liver disease: Any patients with a history of ascites, hepatic encephalopathy, variceal bleeding, jaundice, or CTP>7 points should be excluded.
5. History of treatment with nucleos(t)ide analogues other than lamivudine more than 4 weeks
6. History of immune modulatory drugs (interferon, thymosin-alfa) within 24 weeks of screening
7. Liver transplant patient
8. Patient co-infected with HIV, HCV, or HDV
9. Patient with metabolic or genetic liver disease that may affect serum ALT level
10. Habitual alcohol consumption (>140 g/week for male, >70 g/week for female)
11. Patient not able to stop drugs that may affect ALT or HBV DNA level during study periods (ie. Steroid, immune-suppressants, non-steroidal anti-inflammatory drugs, acetaminophen,)
12. Pregnant or lactating woman
13. Menstruating woman unwilling to use appropriate methods of contraception (ie. Condom, oral contraceptives, tubal ligation)
14. Patient with hepatocellular carcinoma (treated or not treated)
15. Patient with any untreated malignancy
16. Patient with history of malignancy cured within 5 years of screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-05; Primary Completion 2013-12 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
The mean reduction of serum HBV DNA from the baseline at week 52. | up to the end of year 1 (52 weeks)

SECONDARY OUTCOMES:
HBV DNA undetectability(<20 IU/mL) | up to the end of year 1 (52 weeks)
  At the end of year 1 in the two groups, HBV DNA undetectability by real time PCR will be assessed.
mean serum HBV DNA level | up to the end of year 1 (52 weeks)
rate of ALT normalization | up to the end of year 1 (52 weeks)
rates of HBeAg loss | up to the end of year 1 (52 weeks)
rate of HBeAg seroconversion at week 52. | up to the end of year 1 (52 weeks)

OTHER OUTCOMES:
Antiviral resistance rate | up to the end of year 1 (52 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Hyung Joon Yim, M.D, Principal Investigator — Korea University
Locations (1):
- Korea University Ansan Hospital, Ansan, Gyeonggi-do, South Korea